CLINICAL TRIAL: NCT05739097
Title: Prospective Study on Feto-maternal outcoMe In aNemIc womEn : MINNIE Study
Brief Title: Prospective Study on Feto-maternal outcoMe In aNemIc womEn
Acronym: MINNIE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Casa Sollievo della Sofferenza IRCCS (Other)
Collaborators: University of Foggia (Other); University of Bari (Other)
Responsible Party: Sponsor
Other Study IDs: MINNIE, version 12/06/2021
Record Dates: First submitted 2023-01-27; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Anemia; Pregnancy Anemia; Pregnancy Bleeding; Transfusion-dependent Anemia; Transfusion; Embolism, Thrombus; Bleeding; Placenta Diseases
MeSH Terms: conditions — Anemia; Embolism; Thrombosis; Hemorrhage; Placenta Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- non-anemic women: Pregnant women consecutively observed at Ob/Gyn Dept
  Interventions: Diagnostic Test: iron deficiency, coagulation abnormalities
- anemic women: Pregnant women at Ob/Gyn Dept
  Interventions: Diagnostic Test: iron deficiency, coagulation abnormalities
- bleeders: Pregnant women at Ob/Gyn Dept
  Interventions: Diagnostic Test: iron deficiency, coagulation abnormalities

INTERVENTIONS:
Diagnostic Test: iron deficiency, coagulation abnormalities — avoid transfusions, where possible

SUMMARY:
Background Blood transfusions in pregnancy are usually urgent, unpredictable, and occur in otherwise healthy women. There is evidence of increasing rates of maternal red blood cell (RBC) transfusion around childbirth both in Europe and in US. Indeed, they are recorded in approximately 0.4-1.6% of all deliveries. Although obstetric patients use a small proportion of the blood supply overall (3-4%), however over the last years there has been a significant increase (about 30%) in the use of blood and blood products throughout pregnancy. Most available data relate to the peri-partum period, defined as those occurring from 48 hours before delivery onwards.

Anemia in pregnancy is associated with increased maternal mortality and fetal intrauterine growth restriction (IUGR). The risk of these adverse effects is proportional to the severity of anemia; for instance, preterm birth and low birth weight rates are particularly high among women with a hemoglobin below 7 g/dL.

The presence of anemia in at-term pregnant women is a rather frequent and unrecognized risk factor for peri-partum hemorrhage (PPH) transfusion. In a retrospective investigation, we have calculated that almost 20% of at-term pregnant women show iron deficiency anemia. It has been suggested that reduction of RBC transfusion in the context of PPH may decrease maternal mortality and, at the same time, reduce costs.

Patient's Blood Management (PBM) is a well-known strategy based on 1) identification of anemia; 2) reduction of blood loss and 3) reduction of RBC transfusion. In several medical specialties, recommendations based on available evidence highlighted the concept that a restrictive RBC administration is safe and efficacious. Despite the fact that the WHO has recommended PBM early 2010, the majority of hospitals are in need of guidelines to apply PBM in daily practice.

Rationale Anemia is a frequent and often unrecognized hallmark of at-term pregnancies. Systematic collection of data on transfusion practice during pregnancy and post-partum period are scarce.

The application of PBM in obstetrics is expected to improve pregnancy outcome and optimize resources.

Objectives Objectives of the present study are

1. To estimate: frequency of anemia in pregnancy and feto-maternal complications, distribution of haemorrhage aetiologies and transfusion indications.
2. To evaluate associations of these outcomes with gestational age, and transfusion dose.

DETAILED DESCRIPTION:
Design Prospective observational study. All consecutive pregnant women referred from January 1st 2022 to January 30th 2023 to PBM service at University of Foggia and IRCCS "Casa Sollievo della Sofferenza " , who will deliver at Ob/Gyn department in the same Institutions. Investigators will collect baseline clinical characteristics, blood count and all available laboratory parameters. Afterwards, investigators will collect feto-maternal outcomes, included data on possible transfusions.

Estimated Sample size : 2000 pregnant patients.

ELIGIBILITY:
Inclusion criteria:

1. all consecutive pregnant women who will sign the informed consent referred to Ob/Gyn dept. at University of Foggia, University of Bari and IRCCS "Casa Sollievo della Sofferenza " to deliver from January 1st 2022 to January 30th 2023

   Exclusion criteria:
2. Not signed informed consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Investigators will enroll consecutive pregnant women hospitalized for delivery from January 1st 2022 to January 30th 2023 to Ob/Gyn dept. at University of Foggia and IRCCS "Casa Sollievo della Sofferenza " .
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
number of maternal deaths or venous thromboembolisms, hemorrhages | 3 months
  investigators will record maternal deaths; thrombosis; hemorrhage; anemia

SECONDARY OUTCOMES:
number of fetal deaths or intrauterine growth restriction | 3 months
  investigators will record number of fetal deaths and fetal growth restriction;

CONTACTS AND LOCATIONS:
Overall Officials: Elvira Grandone, MD, Principal Investigator — CSS
Locations (2):
- Italy (2):
  - Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia
  - Gabriella Cicerone, Foggia

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2021-06-12): https://cdn.clinicaltrials.gov/large-docs/97/NCT05739097/Prot_000.pdf